CLINICAL TRIAL: NCT05984342
Title: Adjuvant Chemotherapy in Combination With Tislelizumab in Lymph Node-Positive Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Affiliated Cancer Hospital of Shantou University Medical College (Other)
Responsible Party: Principal Investigator, Shao-bin Chen, Professor, Affiliated Cancer Hospital of Shantou University Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023045
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinoma; immunotherapy; chemotherapy; surgery; adjuvant therapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — tislelizumab; 130-nm albumin-bound paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adjuvant Chemotherapy in Combination With Immunotherapy (Experimental): Adjuvant Chemotherapy in Combination With Tislelizumab was used in patients with Lymph Node-Positive Esophageal Squamous Cell Carcinoma after surgery
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Adjuvant Chemotherapy （nab-paclitaxel 260mg/m2 d1 plus Cisplatin 75mg/m2 d1 or 25mg/m2 d1-3) in combination with Tislelizumab (200 mg Q3W)
  Other Names: nab-paclitaxel; Cisplatin

SUMMARY:
Esophageal cancer is one of the most common malignancies in China, and esophageal squamous cell carcinoma (ESCC) is the predominant histological type. Surgical resection is still a standard therapeutic approach for patients with resectable ESCC, but the prognosis is still disappointing. Although neoadjuvant chemoradiotherapy plus surgery is currently recommended for patients with locally advanced ESCC, it is still an infrequently used procedure in China. The efficacy of adjuvant therapy on ESCC is still controversial. Recently, the CheckMate 577 trial showed that adjuvant nivolumab therapy could improve DFS for patients with residual disease after neoadjuvant chemoradiotherapy plus surgery. However, no optimal postoperative adjuvant therapy was recommended for patients with ESCC received upfront surgery. We designed a prospective randomized controlled tial to study whether immunotherapy could be used with chemotherapy after surgery to improve overall survival in these patients. The primary endpoint of the study is disease free survival, with secondary endpoints of overall survival, safety and toxicity, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 70 years
2. Untreated before surgery (e.g. radiotherapy, chemotherapy, target therapy and immunotherapy)
3. Histologically documented squamous cell carcinoma of the thoracic esophagus with positive lymph nodes （T1-3N1-3M0）
4. undergoing radical esophagectomy
5. ECOG (Eastern Cooperative Oncology Group) : 0-1
6. No recurrent disease before adjuvant therapy
7. Normal hemodynamic indices before the recruitment
8. Able to understand this study and have signed informed consent

Exclusion Criteria:

1. previous or concurrent malignancy
2. Interstitial lung disease
3. Requiring systemic treatment with either corticosteroids or other immunosuppressive medications
4. Known or suspected allergy to chemotherapeutic drugs or Tislelizumab
5. Active autoimmune disease
6. Active hepatitis
7. Those whom the investigator considered unsuitable for inclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-02 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
disease-free survival rate | 1 years after surgery
  disease free survival after surgery

SECONDARY OUTCOMES:
Rate of adverse events | within 6 months
  Rate of adverse events according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI- CTCAE v5.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Shantou University Medical College, Shantou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided